CLINICAL TRIAL: NCT02890758
Title: Phase I Trial of Universal Donor NK Cell Therapy in Combination With ALT-803
Brief Title: Phase I Trial of Universal Donor NK Cell Therapy in Combination With ALT803
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brenda Cooper, MD (Other)
Responsible Party: Sponsor-Investigator, Brenda Cooper, MD, Medical Oncology Specialist, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2Z16
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Acute Lymphoblastic Leukemia; Chronic Myeloid Leukemia; Chronic Lymphocytic Leukemia; Non Hodgkin Lymphoma; Hodgkin Lymphoma; Myeloproliferative Syndromes; Plasma Cell Myeloma; Colon Carcinoma; Adenocarcinoma of Rectum; Soft Tissue Sarcoma; Ewing's Sarcoma; Rhabdomyosarcoma
Keywords: Natural Killer Cell; ALT-803
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Colonic Neoplasms; Rectal Neoplasms; Sarcoma; Sarcoma, Ewing; Rhabdomyosarcoma | interventions — Cell Count; ALT-803; Cytokines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cytokine Arm (Experimental): Two infusions of Natural Killer (NK) cells and ALT803
  Interventions: Biological: Natural Killer (NK) Cells; Biological: ALT803
- No Cytokine Arm (Active Comparator): Two infusions of Natural Killer (NK) Cells
  Interventions: Biological: Natural Killer (NK) Cells

INTERVENTIONS:
Biological: Natural Killer (NK) Cells — Dose escalation of Natural Killer (NK) Cells from two infusion of starting at Dose Level 1 (1x10^7 cells/kg), dose Level-1 (1x10^6 cells/kg) if 2 of 6 patients at Level 1 develop DLTs. Escalation to dose level 2 (2.5X10^7) and Dose level 3 (5X10^7) is dependent on DLT
Biological: ALT803 — given at 6mcg/kg weekly for four weeks
  Other Names: Cytokine
  Arms: Cytokine Arm

SUMMARY:
The purpose of this study is to find the number of natural killer (NK) cells from non-HLA matched donors that can be safely infused into patients with cancer. NK cells are a form of lymphocytes that defend against cancer cells. NK cells in cancer patients do not work well to fight cancer. In this study, the NK cells are being donated by healthy individuals without cancer who are not "matched" by human leukocyte antigen (HLA) genes to patients. After receiving these NK cells, patients may also be given a drug called ALT803. ALT803 is a protein that keeps NK cells alive, helps them grow in number and supports their cancer-fighting characteristics. HLA-unmatched NK cell infusion is investigational (experimental) because the process has not approved by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
Primary Objective:

To determine the maximum tolerated dose (MTD) of ex vivo expanded non-HLA matched donor NK cells in combination with ALT-803

Secondary Objectives:

* Describe safety profile / toxicity of combining ALT-803 with NK cell adoptive therapy.
* Determine antitumor activity of allogeneic NK cells with ALT-803 support.
* Determine if a lymphocyte depleting regimen is adequate for preventing early elimination of HLA-mismatched donor NK cells by host T-cells.

Study Design:

This is a phase I study with "3+3" design with three planned dose levels of NK cells and a fixed dose of ALT-803. Three patients will be enrolled sequentially to each dose level, starting with dose level 1. Patients will be segregated to either receive ALT803 as cytokine support after NK cell infusion (starting with same dose level as Level 1) or no cytokine administration. Patients in the arm receiving ALT803 will be either hematologic malignancy patients (Cohort A) or Colon/Soft tissue sarcoma patients (Cohort B). Absence of dose limiting toxicity (DLT) in the DLT assessment period of 28 days must be documented for all patients enrolled a cell dose without ALT803 before the next cohort of patients to receive cytokines at that dose level can be enrolled. Patients can also be enrolled in parallel to the next cell dose level without cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic confirmation of relapsed and or refractory hematologic malignancy, locally advanced or metastatic colon/rectal carcinoma, or refractory and/or relapsed soft tissue sarcomas and have failed at least one standard line of therapy.
* Patients will be eligible if they have either declined standard treatment regimens or if there is no standard approach to curative salvage therapy per National Comprehensive Cancer Network (NCCN) guidelines in the setting of relapsed/refractory disease.
* In addition, patients for whom a potential 29-day delay in treatment will not interfere with the subject's potential therapeutic options can be eligible per the treating physician's discretion.

Malignancies can include:

* Acute myeloid leukemia
* Myelodysplastic syndrome
* Acute lymphoblastic leukemia
* Chronic myeloid leukemia
* Chronic lymphocytic leukemia
* Non Hodgkin Lymphoma
* Hodgkin Lymphoma
* Myeloproliferative syndromes
* Plasma cell myeloma
* Colon/rectal carcinoma
* Soft tissue sarcomas including but not limited to Ewing's sarcoma and Rhabdomyosarcoma

  * Patients must have recovered from acute toxicities of prior chemotherapy or stem cell transplant. Any prior non-hematologic vital organ toxicity (cardiac, pulmonary, hepatic, renal) of previous therapy must have resolved to grade 1 or less.
  * All previous chemotherapy or radiation must be completed at least 3 weeks prior to study entry. Immunologic therapy must be completed at least 3 weeks prior to study entry. Patients with prior stem cell transplant must be greater than 365 days post-transplant.
  * Eastern Cooperative Oncology Group (ECOG) performance status ≤2
  * Organ function criteria (There is no exclusion for the presence of cytopenias),

    * Serum total bilirubin <2 mg/dl (except if known Gilbert syndrome and normal transaminases)
    * Aspartate aminotransferase (AST) (SGOT) < 2.5 X institutional upper limit of normal
    * Alanine aminotransferase (ALT) (SGPT) < 2.5 X institutional upper limit of normal
    * Pulmonary function (DLCO) >40% of the expected value corrected for alveolar volume and hemoglobin
    * Serum Creatinine ≤ 1.5 X institutional upper limit of normal
  * Subjects must have the ability to understand and the willingness to sign a written informed consent document.
  * Women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) 4 weeks prior to study entry and for the duration of study participation. Women of child-bearing age must have documented negative pregnancy test prior to start of lympho-depleting regimen.

Exclusion Criteria:

* Subjects receiving any other investigational agents.
* Subjects for whom a potential 29-day delay in treatment will interfere with the subject's potential therapeutic options.
* Patients with untreated malignant involvement of the central nervous system (CNS) should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Head imaging will be necessary to document absence of CNS involvement in patients with colon/rectal cancer and soft tissue sarcomas. Patients with hematologic malignancies who have undergone treatment for malignant involvement of the CNS must have no evidence of residual disease by imaging or CSF sampling prior to study enrollment.
* History of allergic reactions to chemotherapy agents used in this protocol as part of lymphodepletion regimen (Fludarabine and Cyclophosphamide)
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing active uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with chemotherapeutic agents. In addition, these patients are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Chronic active untreated hepatitis B or C infection.
* Recipients of previous allogeneic transplants who have rash involving more than 10% body surface area attributed to graft versus host disease (GVHD) (> Grade 1 GVHD of skin). Stem cell transplant recipients will be excluded if they are still receiving immunosuppression including steroids for GVHD or have active GVHD in any organ (except for Grade 1 only of skin, not requiring treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
MTD of ex vivo expanded non-HLA matched donor NK cells in combination with ALT-803 | Up to 28 days
  MTD Will be determined by dose limiting toxicity (DLT). The MTD will be defined as the dose level immediately below that at which 2 of 6 subjects experience a dose limiting toxicity.
Number of participants without Graft Versus Host Disease (GVHD) | up to 28 days after beginning treatment
  Measure of safety of natural killer (NK) cells in the absence of HLA matching

SECONDARY OUTCOMES:
Number of patients with hematological response | Up to 12 months after beginning treatment
  Complete Remission (CR): Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0x10^9/L; platelet count >100x10^9/L.
  CR with incomplete recovery (CRi): All CR criteria except residual neutropenia or thrombocytopenia.
  Partial Remission (PR):Hematologic criteria of CR; decrease of bone marrow blast percentage to 5-25%; and decrease of pretreatment bone marrow blast percentage by ≥50%.
  Cytogenetic CR (CRc): Reversion to normal karyotype at the time of morphologic CR.
  Resistant disease (RD): Failure to achieve CR, CRi, or PR. Death in aplasia: Deaths occurring ≥7 days after initial treatment. Death from indeterminate cause: Deaths before completing therapy, or <7 days following completion; or deaths occurring ≥7 days after therapy with no blasts in the blood Relapse: Bone marrow blasts ≥ 5%; or reappearance of blasts in the blood; or development of extramedullary disease
Patients response for radiographically measurable lesions | Up to 12 months after beginning treatment
  * Measurable disease: at least one measurable lesion.
  * Measurable lesions: those that can be measured in at least one dimension as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
  * Non-measurable lesions: all other lesions, including small lesions that are not confirmed and followed by imaging techniques.
  * Baseline documentation of "Target" lesions: all measurable lesions up to a maximum of five lesions per organ and 10 lesions in total. Target lesions should be selected on the basis of their size and their suitability for accurate repeated measurements.
  * Non-target lesions: all other lesions should be identified as non-target lesions. Non-target lesions include measurable lesions that exceed the maximum numbers per organ or total of all involved organs as well as non-measurable lesions.
Patients with malignant lymphoma response | Up to 12 months after beginning treatment
  Lymphoma response of Complete remission, partial remission, relapsed disease, stable disease, progressive disease and best response based on the Journal of Clinical Oncology criteria defined by Cheson in 2014
Patients response for Waldenstrom's macroglobulinemia (WM) | Up to 12 months after beginning treatment
  * Complete response (CR): complete disappearance of disease at and negative serum immunofixation.
  * Partial response (PR): >50% reduction of serum monoclonal protein concentration with >50% reduction of tumor infiltrate and resolution of symptoms attributable to WM.
  * Minor response (MR): > 25% but l<50% reduction of serum monoclonal immunoglobulin M (IgM) determined by protein electrophoresis and no new symptoms or signs of active disease.
  * Stable disease: < 25% reduction and <25% increase of serum monoclonal IgM without progression of adenopathy, organomegaly, cytopenias, or clinically significant symptoms caused by disease and/or signs of WM.
  * Progressive disease: fails to meet criteria for response or stable disease. Progression also requires at least a 25% increase of serum monoclonal protein from the lowest value or worsening of cytopenias, lymphadenopathy, or organomegaly, or appearance of disease-related complications.
Patients response for cutaneous lymphomas | Up to 12 months after beginning treatment
  CR/CCR
  * Complete resolution of skin patches, plaques and tumors (or erythroderma)
  * No evidence of abnormal lymph nodes
  * Absence of circulating Sézary cells
  * No evidence of new tumor (CCR) plus confirmation by skin biopsy (CR) PR
  * ≥50% improvement in the summation of (∆ Skin + ∆ Lymph Node + ∆ Peripheral Blood) with at least ≥30% improvement in ∆ Skin
  * No worsening in Lymph Node or Sézary cells
  * No evidence of new tumors (cutaneous or non-cutaneous)
  Stable Disease at 90 Days (SD90)
  • Fails to meet criteria for PR or CR but absence of new cutaneous or non-cutaneous disease over 90 days
  Progressive Disease (PD)
  * ≥ 50% increase from nadir or baseline in styrylpyridine derivative (SPD) or any node or lesion
  * ≥ 50% increase from nadir in gestational trophoblastic disease (GTD) of any node previously >1cm in shortest diameter
  * Appearance of any new cutaneous or non-cutaneous lesion during or at the end of therapy.
Patients response for multiple myeloma | Up to 12 months after beginning treatment
  Stringent Complete Response (sCR)
  * CR as defined below plus:
    • Normal FLC ratio and Absence of clonal cells in bone marrow CR
  * Negative immunofixation on the serum and urine and:
    * Disappearance of any soft tissue plasmacytomas
    * ≤5% plasma cells in bone marrow Very good partial response (VGPR)
  * Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100mg per 24h PR
  * ≥ 50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥ 90% or to <200 mg per 24h
  * If the serum and urine protein are unmeasurable, ≥ 50% decrease in the difference between involved and uninvolved FLC levels is required
  * If the serum and urine protein are unmeasurable, and serum free light assay is also unmeasurable, ≥ 50% decrease in plasmacells is required SD
  * Not meeting criteria for CR, VGPR, PR, or progressive disease
Patients response for chronic myeloid leukemia (CML) | Up to 12 months after beginning treatment
  Complete hematologic response
  • White blood cell count <10,000/microL with no immature granulocytes and <5 percent basophils on differential, platelet count <450,000/microL, and spleen not palpable.
  Cytogenetic responses
  * Complete cytogenetic response: No Philadelphia chromosome positive cells present.
  * Partial cytogenetic response: 1 to 35 percent Philadelphia chromosome positive cells present.
  * Major cytogenetic response includes patients with complete and partial cytogenetic response (ie, 0 to 35 percent Philadelphia chromosome positive cells present).
  * Minor-minimal cytogenetic response: 36 to 95 percent Philadelphia chromosome positive cells present.
  Molecular response:
  * Complete molecular response: break cluster region - Abelson family kinases (BCR-ABL) transcript nondetectable and nonquantifiable in an assay that has at least 4 to 5 log range.
  * Major molecular response: An at least three log reduction in BCR-ABL transcript levels from baseline.
Patients response for metastatic colon/rectal carcinoma and soft tissue sarcomas | Up to 12 months after beginning treatment
  Complete Response: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm (the sum may not be "0" if there are target nodes). Partial Response: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions may be considered progression).
  Stable Disease: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
Average duration of response | Up to 12 months after beginning treatment
  The duration of overall response is measured from the time of NK Cell infusion until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Average duration of Overall Survival | Up to 12 months after beginning treatment
  Overall survival is measured from the date of first infusion of NK cells to the date of death from any cause; patients not known to have died at last follow up are censored on the date they were last known to be alive.
Average duration of relapse free survival | Up to 12 months after beginning treatment
  Only those patients achieving complete response (CR) or complete response with incomplete recovery (CRI). It is measured from the date of infusion of NK cells until the date of relapse or death from any cause; patients not known to have relapsed or died at last follow up are censored on the date they were last examined.
in vivo Natural Killer (NK) levels | up to 28 days after beginning treatment
  Measurement of in vivo NK cell levels following cell product infusion will be done on peripheral blood by flow cytometry (CD3- CD56+ positive cells). This will be done on peripheral blood samples of patients. Measurement of successful donor NK cell persistence (absence of cell product rejection) will be defined as measurement of >100 NK cell/µL

CONTACTS AND LOCATIONS:
Overall Officials: David Wald, MD, PhD, Study Director — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States